CLINICAL TRIAL: NCT05235945
Title: The Effect of a Preoperative Exercise Programme on Cardiorespiratory Fitness, Resting Metabolic Rate and Autonomic Control in Patients With Severe Obesity Awaiting Bariatric Surgery
Brief Title: The Effect of Exercise in Patients Awaiting Bariatric Surgery
Acronym: BariPrehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 130811; 273319 (Registry Identifier: IRAS); 21/EM/0230 (Other: HRA and Health and Care Research Wales (HCRW))
Record Dates: First submitted 2022-01-12; First posted 2022-02-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery Candidate; Obesity
Keywords: exercise; fitness; pre-operative; prehabilitation; bariatric; obesity; surgery
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online exercise intervention (Experimental): A four-week preoperative physical activity intervention, involving a combination of supervised and unsupervised (live or pre-recorded), online exercise sessions. These sessions will be designed to meet the National physical activity guidelines (2020) of at least 150 minutes of low-moderate or 75 minutes of vigorous physical activity per week (or a combination of the two). The intervention will involve moderate intensity activities that aim to increase or maintain muscle strength (resistance training) as well as short bouts of vigorous aerobic exercise, using major muscle groups in the lower and upper body.
  Interventions: Behavioral: Online exercise intervention
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Online exercise intervention — Described in arm descriptions
  Arms: Online exercise intervention

SUMMARY:
The aim of this project is to understand the impact of a four week preoperative exercise programme on fitness and metabolic rate and weight before surgery.

A multi-site randomised trial sponsored by UCL, recruiting patients awaiting bariatric surgery for obesity at University College London Hospital (UCLH), Whittington Health NHS Trust, or Homerton University Hospital NHS Foundation Trust.

The investigators will measure fitness, metabolic rate, body weight/composition and grip strength in all participants, before and after a four-week supervised physical activity intervention. The investigators will also interview participants about their participation in the study in regard to the planning of future studies.

DETAILED DESCRIPTION:
The aim of this project is to understand the impact of a structured personalised 4-week exercise programme on resting fitness and metabolic rate in patients awaiting bariatric surgery for obesity. The hypothesis is that patients awaiting bariatric surgery who undertake a preoperative exercise programme will experience attenuated changes in functional capacity (fitness) and metabolic rate compared with usual care (no exercise programme) along with alterations in autonomic control.

The investigators propose a randomised controlled trial that will recruit 48 patients with obesity scheduled for bariatric surgery at UCLH, Whittington Health NHS Trust, and Homerton University Hospital NHS Foundation Trust. Participants will be randomly assigned to either usual care (exercise advice only) or combination exercise intervention group, during a four-week lead up to surgery, on a 1:1 basis.

Participants randomised to the intervention group will participate in 7 physiologist-led exercise sessions online and also be instructed to complete 7 self-led 30-minute exercise sessions over the four-week intervention period. This equates to a total of 14 exercise sessions across the four-week (28 day) intervention. Additionally, participants will be encouraged to be physically active on as many days as possible, in bouts of 10-minutes or more. The programme is designed to meet the National Physical Activity Guidelines of at least 150 minutes of low-moderate or 75 minutes of vigorous PA per week, or a combination of the two.

The investigators will measure physical fitness, metabolic rate, and how the heart responds to hormonal changes (the sympathetic nervous system) in all participants, before and after the four-week study period. The investigators will also interview participants about their participation in the study in regard to the planning of future studies.

Baseline data collection will occur at least six weeks prior to surgery as detailed below. Both groups will be invited to attend follow-up assessment at 4 weeks where they will undergo the same series of tests. The total duration of participation will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18 and above.
2. Patients enrolled in the UCLH, Homerton or Whittington Hospitals bariatric surgery program with BMI > 30 kg/m2
3. ≤5 % variation in body weight over preceding 3 months.
4. Willing and able to comply with the trial protocol.
5. Willing and able to provide written informed consent
6. Male or Female

Exclusion Criteria:

1. Pregnant or lactating mothers.
2. Weight over 180 kg (due to weight restrictions of equipment used).
3. Current use of betablockade.
4. Concurrent participation in other clinical intervention trial.
5. Clinically significant medical co-morbidities (e.g. uncontrolled hypertension, unstable cardiovascular disease) that could place at risk of an adverse response to exercise.
6. History of atrial fibrillation, unstable angina, acute coronary syndrome, congestive heart failure New York Heart Association class III-IV within the preceding 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fitness (VO2 in ml/kg/min) | 4 weeks
  VO2 (at anaerobic threshold (AT) and peak exercise) using gas-analysed cardiopulmonary exercise testing.

SECONDARY OUTCOMES:
Resting metabolic rate (VO2 in ml/kg/min) | 4 weeks
  Energy expenditure at rest, collected using respiratory gas-analysis via metabolic cart.
Maximal grip strength (kg) | 4 weeks
  Hand grip dynamometry, best of three repeat measures on each hand (left and right)
Body mass (kg) | 4 weeks
  Body mass in kilograms using body weight scales.
Autonomic control (heart-rate variability) | 4 weeks
  Heart-rate variability measured via electrocardiogram (ECG), assessing the variability between heart beats at rest, resting heart-rate, and exercise heart-rate response
Participant satisfaction feedback | 4 weeks
  Participants satisfaction/acceptability of the mode of delivery and content of the intervention will be collected via semi-structured interviews. Participants will be asked how much they liked specific aspects of the program, and will answer using a 5-point Likert scale. They will also be asked to provide general feedback, and answers related to behaviour change using open-ended questions.
Body composition (%FM, %FFM) | 4 weeks
  Percent fat mass and percent fat-free mass using bioelectric impedance analysis (BIA)
Physical activity patterns | 7 days
  7-day physical activity patterns (sedentary time, low, moderate and vigorous physical activity) measured using accelerometer data

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Durey, Principal Investigator — UCL, UniSA and UNSW
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Summary format only, Access to IPD will be reviewed on a case-by-case basis following requests.

REFERENCES:
- [Result] Durey BJ, Fritche D, Martin DS, Best LMJ. The Effect of Pre-operative Exercise Intervention on Patient Outcomes Following Bariatric Surgery: a Systematic Review and Meta-analysis. Obes Surg. 2022 Jan;32(1):160-169. doi: 10.1007/s11695-021-05743-w. Epub 2021 Oct 20. PMID 34671929
- [Result] Sardeli AV, Komatsu TR, Mori MA, Gaspari AF, Chacon-Mikahil MPT. Resistance Training Prevents Muscle Loss Induced by Caloric Restriction in Obese Elderly Individuals: A Systematic Review and Meta-Analysis. Nutrients. 2018 Mar 29;10(4):423. doi: 10.3390/nu10040423. PMID 29596307
- [Derived] Durey BJ, Coates AM, Davison K, Tarca B, Mok J, Parmar CD, Fernandez-Munoz N, Burton K, Tetlow N, Dewar AL, Adeleke MO, Lugg Z, Colbert J, Martin DS. Evaluating the Impact of Telehealth Exercise Prehabilitation on Cardiometabolic Health in Bariatric Surgery Candidates: Protocol for the BARI-Prehab Randomized Controlled Trial. JMIR Res Protoc. 2025 Nov 13;14:e77538. doi: 10.2196/77538. PMID 41232096